CLINICAL TRIAL: NCT04220437
Title: Identification of Neoatherosclerosis in In-stent Restenosis Patients Based on Artifical Intelligence
Brief Title: Identification of Neoatherosclerosis in ISR Patients Based on Artifical Intelligence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Professor, Chinese PLA General Hospital
Other Study IDs: AI-301-ISR
Record Dates: First submitted 2019-12-21; First posted 2020-01-07 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: In-stent Restenosis; Neo-atherosclerosis; Retrospective
Keywords: Neoatherosclerosis; in-stent restenosis; Optical Coherence Tomography; angiography; artificial intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAG and OCT group: Images of CAG and OCT patients obtained from ISR patients were retrospectively collected and analyzed.
  Interventions: Other: no interventin

INTERVENTIONS:
Other: no interventin — Our stusy analysed the images obtained from ISR patients, no extra intervention was given based on this study.

SUMMARY:
Based on the large population of patients, in-stent restenosis (ISR) is still an important problem in the field of cardiovascular disease. How to reduce the incidence of ISR and the treatment of ISR has become the focus and hot spot. The 2018 ESC Guidelines for Cardiovascular Intervention recommends treatment of ISR under the guidance of intravascular ultrasound (IVUS), or optical coherent tomography (OCT). Circulation published a new Waksman ISR classification based on mechanisms and components of the restenosis tissue, which provides guidance for treatment strategy. Because of its good resolution, OCT makes it more accurate to distinguish the components of vascular tissue, thus providing a decision-making basis for interventional therapy. OCT examination can obtain the characteristics of the ISR more precisely. Neoatherosclerosis (NA), is one of the ISR types and accounts for more stent failure and target lesion failure than other types. Identification NA is important for decision-making of interventional therapy. However, the acquisition and analysis of OCT images not only need the digital angiography machine (DSA) equipped with the majority of hospitals, but also need professional OCT imaging equipment and technicians. Patients with severely CKD cannot bear OCT examination because of the large amount of contrast agent. OCT catheter is more than ten times the price of the CAG catheter. Therefore, identification of NA by the use of artificial intelligence (AI) is of significance to set therapeutic strategy for ISR patients, especially in patients with CKD. Our study retrospectively analyzed CAG images and OCT images of ISR patients obtained from Jan 1st,2015 to Oct 31st,2020. Identify NA by analyzing OCT images, build up U-net and V-net to analyze the CAG and OCT images, and finally build up an identification system of NA based on CAG images by AI. This study has been approved by Ethics Committee of Chinese PLA General Hospital (S2018-033-01)

DETAILED DESCRIPTION:
Drug Eluting Stents (DES) reduce the rate of in-stent restenosis (ISR) to 3.6-10%. Based on the large population of patients, ISR is still an important problem in the field of cardiovascular disease. How to reduce the incidence of ISR and the treatment of ISR has become the focus and hot spot. The 2018 ESC Guidelines for Cardiovascular Intervention recommends treatment of ISR under the guidance of intravascular ultrasound (IVUS), or optical coherent tomography (OCT). The European Expert Consensus on Intravascular Imaging, published in 2018, recommends finding the underlying mechanisms of ISR through intravascular imaging guidance (IVUS or OCT), and determining therapeutic strategies based on the mechanisms. Circulation published a new Waksman ISR classification based on mechanisms and components of the restenosis tissue, which provides guidance of treatment strategy. The use of intravascular imaging to identify and classify the types and mechanisms is very important for ISR treatment strategy. Because of its good resolution, OCT makes it more accurate to distinguish the components of vascular tissue, thus providing a decision-making basis for interventional therapy. OCT examination can obtain the characteristics of ISR more precisely. Neoatherosclerosis (NA), is one of the ISR types and accounts for more stent failure and target lesion failure than other types. Identification of NA is important for decision-making of interventional therapy. However, the acquisition and analysis of OCT images not only need the digital angiography machine (DSA) equipped with the majority of hospitals, but also need professional OCT imaging equipment and technicians. Patients with severely CKD cannot bear OCT examination because of the large amount of contrast agent. OCT catheter is more than ten times the price of the CAG catheter. Therefore, identification of NA by the use of artificial intelligence (AI) is of significance to set therapeutic strategy for ISR patients, especially in patients with CKD. Our study retrospectively analyzed CAG images and OCT images of ISR patients obtained from Jan 1st,2015 to Jan 31st,2020. Offline OCT analysis was performed using dedicated software (Light Lab Imaging Inc, Westford, MA). All images were analyzed at every frame in the stents by 2 independent investigators, who were blinded to the angiographic and clinical findings. Identify NA by analyzing OCT images, build up U-net and V-net to analyze the CAG and OCT images, and finally build up an identification system of NA based on CAG images by AI. This study has been approved by Ethics Committee of Chinese PLA General Hospital (S2018-033-01)

ELIGIBILITY:
Inclusion Criteria:

- all gender

18ys old to 80ys old

diagnosed of in-stent restenosis based on CAG

both CAG images and OCT images were obtained in the same patient on the same day

Exclusion Criteria:

* CAG images and OCT images were not obtained on the same day in the same patient

low quality in CAG images

low qualitiy in OCT images

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients were enrolled
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-02-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
The identification of NA | through the study completion, an average of 3 years
  a neointima containing a diffuse border and a signal-poor region, with the struts underneath invisible because of the marked signal attenuation
neovascularizaion | through the study completion, an average of 3 years
  diameter 50-300um, cavity in the stent area, not connected with the vasular
ISR segment in the CAG images | through the study completion, an average of 3 years
  the segement in the stent area or within 5mm beside the stent,diameter stenosis rate>50%
lipid-core arc | through the study completion, an average of 3 years
  To quantify the circumferential extent of NA, the lipid-core arc was measured at a 0.2-mm interval throughout the segments showing NA.
Thin-cap fibroatheroma-like neointima | through the study completion, an average of 3 years
  defined as a neointima characterized by a fibrous cap thickness at the thinnest part of <65 μm and an angle of lipid-laden neointima of >180 degrees
macrophage arc | through the study completion, an average of 3 years
  measured at 0.2-mm intervals and divided into 5 groups: grade 0, no macrophages; grade 1, localized macrophage accumulation, <30 degrees; grade 2, clustered accumulation, ≥30 and <90 degrees; grade 3, clustered accumulation, ≥90 and <270 degrees; and grade 4, clustered accumulation, ≥270 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, M.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- The General Hospital of PLA, Beijing, China

IPD SHARING:
Plan to Share IPD: No